CLINICAL TRIAL: NCT05051787
Title: Evaluation of Amoxicillin Diffusion in Breast Milk According to a Population Pharmacokinetic Approach.
Brief Title: Evaluation of Amoxicillin Diffusion in Breast Milk According to a Population Pharmacokinetic Approach (CONCEPTION-AMOX)
Acronym: CONCEPTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/21/0217
Record Dates: First submitted 2021-07-02; First posted 2021-09-21 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Breast Feeding, Exclusive
Keywords: amoxicillin; population pharmacokinetic model
MeSH Terms: conditions — Breast Feeding | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breastfeeding women (Experimental): Mothers over 18, treated with amoxicillin alone or associated with clavulanic acid for at least 2 days, breastfeeding their child.
  Interventions: Biological: Blood and milk samples

INTERVENTIONS:
Biological: Blood and milk samples — 2 types of samples will be taken over the same time slots in breastfeeding mothers treated with amoxicillin for at least 2 days:
  * 3 breast milk collections of about 20 ml each made using an electric breast pump provided to the participant.
  * 3 blood samples of approximately 5 ml each.

SUMMARY:
Based on plasma and milk concentrations, a PopPK model will be performed (i) to document the average and individual exposure to amoxicillin in milk, (ii) to identify the factors explaining the inter-individual pharmacokinetic variability and (iii) to determine the daily dose ingested by the infant and its variability for different dosage regimens applied to the mother. The secondary objectives are to monitor (i) predefined adverse reactions in infants and (ii) the impact on milk production.

DETAILED DESCRIPTION:
This study will complement the clinical data on amoxicillin in breastfed new-borns considering that current knowledge in terms of authorized drugs use during breastfeeding is not sufficient to guarantee the child absence of exposure, even minimal. As a consequence, this lack of certainties leads to premature discontinuation of breastfeeding, well known to be beneficial for the breastfed new-borns. Amoxicillin, prescribed alone or with clavulanic acid at 2 to 3g per day for 7 days, including in lactating women, is mainly used to treat β-hemolytic strep throat, infections of the genitourinary tract as well as ear, nose and throat infections.

ELIGIBILITY:
Inclusion Criteria:

* Mothers over 18 years, treated by amoxicillin for at least 2 days who breastfeed their child, - Participation requires that breastfeeding is already well established (i.e., at least 2 weeks after giving birth in order to sample mature milk) and that the infant is over 4 weeks old,
* Affiliation to the social security scheme or equivalent,
* Ability to understand and willingness to sign a written Informed Consent document.

Exclusion Criteria:

* Mothers under 18 years old,
* Infants born prematurely (i.e., gestational age under 34 weeks) or requiring appropriate medical supervision or support from a team of social workers,
* Mothers who gave birth to twins,
* Inability to communicate due to language problems for the mother,
* Patient subject to a legal protection order (curatorship or tutorship).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Concentration-time profile of amoxicillin in milk | At the time of samplings (day 0)
Concentration-time profile of amoxicillin in plasma | At the time of samplings (day 0)

SECONDARY OUTCOMES:
Occurrence of predefined side effects in infants during the breastfeeding period. | At the time of samplings (day 0) and a week later (day 7)
  Occurrence of diarrhoea, nausea, vomiting, feeding difficulties, skin rashes, urticaria and candidiasis will be monitored using a form on the infant's health status and breastmilk production will be completed by the mother/parent at the time of samplings and a week later.
Impact of mother's drug consumption on breast milk production. | At the time of samplings (day 0) and a week later (day 7)
  A form on breastmilk production will be completed by the mother/parent at the time of samplings and a week later

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Gandia, MD, Study Chair — University Hospital, Toulouse
Locations (2):
- France (2):
  - APHP Hôpital Necker, Lactarium Régional d'Ile de France, Paris
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No